CLINICAL TRIAL: NCT00005723
Title: Worksite Issues in Organizational Health Promotion (Take Heart)
Status: Completed | Type: Observational
Sponsor: Oregon Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4932; R01HL045548 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the impact of organizational-level health promotion activities and worksite characteristics on employee dietary and smoking behaviors.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Based upon the organizational literature on adoption and institutionalization of innovative practices, a disseminable intervention protocol and materials (e.g., a guidebook for worksite health promotion steering committees) was developed. This intervention was evaluated in a randomized control trial comparing 13 treatment worksites to 13 delayed-treatment worksites on organizational health promotion practices (policies/environmental control, incentive programs, skills training activities, maintenance activities); employee smoking cessation and saturated fat consumption; and employee cholesterol levels. Following a two-year assessment, worksites in the delayed-treatment condition received a version of the intervention requiring less interventionist time. The effects of this streamlined intervention in these worksites were evaluated relative relative to a third group of 13 quasi-experimental comparison worksites that entered the study at that time.

The study also evaluated the impact of organization characteristics and health promotion activities on employees at various stages of health related behavior change (awareness, intention to change, behavior change attempt, maintenance of behavior change). Process measures assessing program implementation and cost-effectiveness data were collected. Finally, the long-term intervention effects (3-4 years following initial intervention) on organizational health promotion practices, employee dietary and smoking behaviors, and cholesterol levels were assessed. In summary, this five year project provided both a) knowledge about how to implement worksite health promotion interventions to promote employee ownership and maintenance, and b) disseminable intervention products (e.g., protocols and employee steering committee guidebooks).

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-01; Primary Completion 1996-01 (Actual); Study Completion 1996-09 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Glasgow RE, Terborg JR, Hollis JF, Severson HH, Fisher KJ, Boles SM, Pettigrew EL, Foster LS, Strycker LA, Bischoff S. Modifying dietary and tobacco use patterns in the worksite: the Take Heart Project. Health Educ Q. 1994 Spring;21(1):69-82. doi: 10.1177/109019819402100108. PMID 8188494
- [Background] Glasgow RE, McCaul KD, Fisher KJ. Participation in worksite health promotion: a critique of the literature and recommendations for future practice. Health Educ Q. 1993 Fall;20(3):391-408. doi: 10.1177/109019819302000309. PMID 8307762
- [Background] Glasgow RE, Terborg JR, Strycker LA, Boles SM, Hollis JF. Take Heart II: replication of a worksite health promotion trial. J Behav Med. 1997 Apr;20(2):143-61. doi: 10.1023/a:1025578627362. PMID 9144037
- [Background] Glasgow RE, Perry JD, Toobert DJ, Hollis JF. Brief assessments of dietary behavior in field settings. Addict Behav. 1996 Mar-Apr;21(2):239-47. doi: 10.1016/0306-4603(95)00056-9. PMID 8730527
- [Background] Glasgow RE, Terborg JR, Hollis JF, Severson HH, Boles SM. Take heart: results from the initial phase of a work-site wellness program. Am J Public Health. 1995 Feb;85(2):209-16. doi: 10.2105/ajph.85.2.209. PMID 7856780